CLINICAL TRIAL: NCT06993558
Title: Analysis of Safety and Tissue Interaction of Injectable and Energy-based Biosmulators.
Acronym: Biostimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Lynhda Nguyen, Dr.med. Lynhda Nguyen, Universitätsklinikum Hamburg-Eppendorf
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-101412-BO-ff; University Hamburg Eppendorf (Other: Medicine Faculty - Clinic and Polyclinic for Dermatology and Venerology)
Record Dates: First submitted 2025-05-19; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: This Study Aims to Evaluate the Safety Profile and Tissue Changes After Biostimulatory Treatments to the Face in Healthy Volunteers
Keywords: Ultrasound; Biostimulation; Poly-L-Lactic-Acid; Calcium-Hydroxylapatit; Radio Frequency Microneedling
MeSH Terms: interventions — poly(lactide); New-Fill; Injections; Durapatite

STUDY DESIGN:
Intervention Model Description: Healthy patients scheduled for biostimulatory treatment (one of three different modalities) at the outpatient clinic will be enrolled in the study. Upon completion of the treatment protocol, participants will undergo a series of follow-up visits. These follow-ups will include standardized 3D photographic documentation, ultrasound assessments, as well as both patient-reported outcome measures and physician-administered evaluations/questionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (3):
- Injectable Biostimulator 1 (Experimental): Injection to the face with a blunt canula
  Interventions: Procedure: Poly-L-Lactic Acid (Sculptra) injection
- Injectable Biostimulator 2 (Experimental): Will be injected to the face with blunt canula
  Interventions: Procedure: Calcium Hydroxyapatite
- Energy-based Biostimulator (Experimental): 1-3 Treatments with 6-8 weeks of intervall
  Interventions: Procedure: Radiofrequency Microneedling

INTERVENTIONS:
Procedure: Poly-L-Lactic Acid (Sculptra) injection — 1 to 2 sessions at intervals of 4 to 6 weeks are planned with PLLA (Sculptra®, Galderma Laboratories). PLLA will be injected into the face or neck region using a blunt cannula. For reconstitution, 7 ml of saline solution and 1 ml of 1 % lidocaine will be used. 5 minutes of massaging for 5 times a day are recommended.
  Arms: Injectable Biostimulator 1
Procedure: Calcium Hydroxyapatite — For CaHA treatment (Radiesse®, Merz Pharma; HarmonyCa®, Allergan), 1 session is planned. The face (cheeks, jawline) or neck will be augmented using a blunt cannula, either diluted (Radiesse® 1:0.2 - 1:2) or undiluted (HarmonyCA®) depending on the product and the region being treated.
  Arms: Injectable Biostimulator 2
Procedure: Radiofrequency Microneedling — For RFMN treatment (Genius®, Lutronic Medical Systems), 1 to 3 sessions at intervals of 6 to 8 weeks are planned. Prior to treatment, subjects were given topical anesthesia (23% lidocaine, 3.5% tetracaine) under occlusion for at least 1.5 hours. The face will be treated with an RFMN system, using parameters adjusted for each anatomical location. Each region received three passes with 50 - 70 % overlap, starting with the longest needle setting. A minimum total energy of 1000 J will be aimed. Treatment will be performed using forced cooled air (Cryo6, Zimmer Aesthe cDivision).
  Arms: Energy-based Biostimulator

SUMMARY:
The goal of this clinical trial is to analyse tissue changes in the pre-auricular region after injectable (Poly-L-Lactic-Acid/Calcium-Hydroxylapatit/ and energy-based (Radiofrequency Microneedling) biostimulatory interventions in healthy volunteers. The main questions it aims to answer are:

How is the Safety Profile of Biostimulatory Treatments? How are the Tissue Interactions after Biostiomulatory Treatments?

Participants will:

* Recieve one of 3 possible biostumulatory treatments (PLLA/CAHA/RFM)
* Attend 5 follow-up appointments after treatment for checkups, surveillance and examinations.

DETAILED DESCRIPTION:
Patients undergoing biostimulatory treatments will be invited to participate in this study involving photographic evaluations and ultrasound imaging. Following detailed oral and written explanations, patients will provide informed consent.

Participants will be assigned to one of three treatment groups:

1. PLLA (Sculptra®, Sinclair Pharmaceuticals)
2. CaHA (Radiesse®, Merz Pharma; HarmonyCa®, Allergan)
3. RFMN (Genius®, Lutronic Medical Systems)

Treatment Protocols:

* PLLA: 1-3 sessions at intervals of 4-6 weeks
* CaHA: Single session
* RFMN: 1-3 sessions at intervals of 6-8 weeks

These interventions will follow routine clinical protocols, with more frequent follow-ups involving photography and ultrasound imaging as part of the study.

Follow-Up Assessments

Patients will undergo follow-up evaluations at 5 defined time points after treatment:

1. 6 weeks
2. 6 months
3. 12 months 4.18 months

5. 24 months

ELIGIBILITY:
-Inclusion Criteria:

Men and women aged 30 years and older

Good general health, no relevant pre-existing conditions

Patients planning to undergo CaHa, PLLA, or RFMN treatment as part of routine care due to skin laxity or volume loss

Cognitive ability and willingness to provide informed consent

Willingness and ability to attend follow-up visits

-Exclusion Criteria:

Age under 30 years

Pregnant or breastfeeding individuals

Significant open wounds or lesions in the treatment area

Metallic implants in the treatment area

Psychiatric disorders (psychosis, body dysmorphic disorders)

Missing informed consent and/or data privacy declarations

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-22 (Actual); Primary Completion 2026-03-22 (Estimated); Study Completion 2026-09-22 (Estimated)

PRIMARY OUTCOMES:
Inflammatory Reaction | From enrollment to the end of treatment at 6-8 week
  The effectiveness of biostimulatory treatments relies on inducing a localized inflammatory response. Ultrasound and optical coherence tomography (OCT) can be used to assess vascular dynamics and edema, serving as objective markers of inflammation.
Analysis of Injected Biostimulator-Deposits | From enrollment to the end of treatment at 6 -8 week
  Injected deposits: In the CaHa and PLLA treatment groups, deposits will be visualized via sonographic imaging, a 3-distance Volume measurement will be performed
Tissue Interaction | From enrollment to the end of treatment at 6-8 weeks
  Characterized through ultrasound and OCT, focusing on the visualization of the epidermis, dermis, superficial fat layer, fibrous layer (fascia/superficial musculoaponeurotic system), deep fat layer, and periosteum.
Adverse Events | From enrollment to the end of treatment at 6-8 week
  If AEs occur, they will be documented with photos, ultrasound, and OCT, with appropriate treatment provided.

SECONDARY OUTCOMES:
Clinical Outcome | From enrollment to the end of treatment at 6-8 week
  Assessed using the Physician and Subject Global Aesthetic Improvement Scale (PGAIS, SGAIS) based on standardized photo documentation.
Patient Satisfaction | From enrollment to the end of treatment at 6-8 week
  Measured using a five-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jair Mauricio Ceron Bohorquez, M.D., Principal Investigator — Medical Contour
Locations (1):
- University Hospital Hamburg Eppendorf, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD) may not be shared due to concerns about participant privacy and data protection regulations, limitations in the original informed consent, intellectual property or commercial interests, and the significant resources required to prepare and anonymize the data. Additionally, ethical considerations and institutional or regulatory policies may further restrict data sharing to ensure participant confidentiality and prevent potential misuse.

REFERENCES:
- [Background] Wortsman X, Quezada N, Penaloza O, Cavallieri F, Schelke L, Velthuis P. Ultrasonographic Patterns of Calcium Hydroxyapatite According to Dilution and Mix With Hyaluronic Acid. J Ultrasound Med. 2023 Sep;42(9):2065-2072. doi: 10.1002/jum.16226. Epub 2023 Mar 27. PMID 36972372
- [Background] Velthuis PJ, Jansen O, Schelke LW, Moon HJ, Kadouch J, Ascher B, Cotofana S. A Guide to Doppler Ultrasound Analysis of the Face in Cosmetic Medicine. Part 2: Vascular Mapping. Aesthet Surg J. 2021 Oct 15;41(11):NP1633-NP1644. doi: 10.1093/asj/sjaa411. PMID 33954749
- [Background] Velthuis PJ, Jansen O, Schelke LW, Moon HJ, Kadouch J, Ascher B, Cotofana S. A Guide to Doppler Ultrasound Analysis of the Face in Cosmetic Medicine. Part 1: Standard Positions. Aesthet Surg J. 2021 Oct 15;41(11):NP1621-NP1632. doi: 10.1093/asj/sjaa410. PMID 33954581
- [Background] Wortsman X, Alfageme F, Roustan G, Arias-Santiago S, Martorell A, Catalano O, Scotto di Santolo M, Zarchi K, Bouer M, Gonzalez C, Bard R, Mandava A, Gaitini D. Guidelines for Performing Dermatologic Ultrasound Examinations by the DERMUS Group. J Ultrasound Med. 2016 Mar;35(3):577-80. doi: 10.7863/ultra.15.06046. Epub 2016 Feb 17. PMID 26887446
- [Background] Kyriazidis I, Spyropoulou GA, Zambacos G, Tagka A, Rakhorst HA, Gasteratos K, Berner JE, Mandrekas A. Adverse Events Associated with Hyaluronic Acid Filler Injection for Non-surgical Facial Aesthetics: A Systematic Review of High Level of Evidence Studies. Aesthetic Plast Surg. 2024 Feb;48(4):719-741. doi: 10.1007/s00266-023-03465-1. Epub 2023 Aug 10. PMID 37563436
- [Background] Pavicic T. Complete biodegradable nature of calcium hydroxylapatite after injection for malar enhancement: an MRI study. Clin Cosmet Investig Dermatol. 2015 Feb 9;8:19-25. doi: 10.2147/CCID.S72878. eCollection 2015. PMID 25709485
- [Background] Amselem M. Radiesse((R)): a novel rejuvenation treatment for the upper arms. Clin Cosmet Investig Dermatol. 2015 Dec 29;9:9-14. doi: 10.2147/CCID.S93137. eCollection 2016. PMID 26766918
- [Background] Yutskovskaya Y, Kogan E, Leshunov E. A randomized, split-face, histomorphologic study comparing a volumetric calcium hydroxylapatite and a hyaluronic acid-based dermal filler. J Drugs Dermatol. 2014 Sep;13(9):1047-52. PMID 25226004
- See also: American Society of Plastic Surgeons Reveals 2022's Most Sought-After Procedures — https://www.prnewswire.com/news-releases/american-society-of-plastic-surgeons-reveals-2022s-most-sought-after-procedures-301938919.html